CLINICAL TRIAL: NCT04258644
Title: Efficacy and Safety of Camrelizumab in Combination With Apatinib Mesylate, Paclitaxel-albumin and S-1 for Translational Treatment of Gastric Cancer
Brief Title: Camrelizumab in Combination With Apatinib Mesylate, Paclitaxel-albumin and S-1 for Translational Treatment of Gastric Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beijing Friendship Hospital (Other)
Responsible Party: Principal Investigator, Zhongtao Zhang, Professor, Beijing Friendship Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BFH-CamrelizumabCombo4
Record Dates: First submitted 2020-02-05; First posted 2020-02-06 (Actual); Last update posted 2020-02-06 (Actual); Status verified 2020-02

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Camrelizumab+Apatinib+Paclitaxel-albumin+S-1 (Experimental): Camrelizumab：D1, 200 mg ivgtt Apatinib Mesylate：D1~21, 250 mg, po qd Paclitaxel-albumin：D1&D8, 100～120 mg/m2 S-1：D1~14, 60mg bid
  Interventions: Drug: Camrelizumab+Apatinib+Paclitaxel-albumin+S-1

INTERVENTIONS:
Drug: Camrelizumab+Apatinib+Paclitaxel-albumin+S-1 — Combination therapy of 4 drugs, 21 days for one cycle.

SUMMARY:
This is an interventional clinical trial to assess the efficacy and safety of camrelizumab in combination with apatinib mesylate, paclitaxel-albumin and S-1 for translational treatment of gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

1. age:18～70; expected survival>3 months
2. pathologically diagnosed gastric cancer or esophageal-gastric-junction cancer, being predominantly adenocarcinoma
3. no previous treatment of anti-cancer drugs
4. ECOG score 0~2
5. CT/MRI/PET-CT diagnosed as unresectable
6. no disfunction of major organs
7. lab results satisfy the following criteria:

   * Hb≥90g/L
   * WBC≥3.5×109/L
   * Neutrophil≥1.5×109/L
   * Plt≥100×109/L
   * ALT、AST≤2.5 upper limit (≤5 upper limit for patients with liver metastasis)
   * Tbil≤1.5 upper limit
   * serum creatinine≤1.5 upper limit

7.women at child-bearing age must be tested negative within 7 days before inclusion, and must be willing to take contraception measures during treatment and within 12 weeks after last dose of treatment; men must be sterilized or willing to take contraception measures during treatment and within 12 weeks after last dose of treatment 8.willing to join this research with hand-signed written Informed consent 9.good compliance for follow-up

Exclusion Criteria:

1. patients with positive HER-2 test
2. with conditions that affect the absorption of oral drugs, such as inability to swallow, nausea and vomiting, chronic diarrhea and intestinal obstruction
3. allergic to carrizumab for injection, apatinib mesylate, paclitaxel for injection (albumin binding type) and tS-1 or relevant drug excipients; allergic to any other monoclonal antibodies; cannot tolerate radiation toxicity;
4. with active autoimmune disease or autoimmune disease history, such as interstitial pneumonia, uveitis, enteritis, hepatitis, hypophysitis, vasculitis, myocarditis, nephritis, hyperthyroidism, hypothyroidism (can be included after hormone replacement therapy); patients with complete remission of childhood asthma and require no intervention can be included, whereas those who need medical intervention with bronchodilator cannot be included
5. with congenital or acquired immune defects, such as human immunodeficiency virus (HIV) infection, active hepatitis B (HBV DNA ≥ 500 IU / ml), hepatitis C (HCV antibody positive, and HCV-RNA higher than the lower detection limit of the analysis method) or combined hepatitis B and hepatitis C co infection
6. immunosuppressive drugs were used within 14 days before the first use of the study drug, excluding nasal spray and inhaled corticosteroids or systemic steroids in physiological dose (i.e. no more than 10 mg / day of prednisolone or other corticosteroids for equivalent amount);
7. inoculated live attenuated vaccine within 4 weeks before the first administration or during the study period
8. severe infection (requiring intravenous drip of antibiotics, antifungal or antiviral drugs) within 4 weeks before the first administration, or fever> 38.5° C of unknown cause during screening / before the first administration
9. known history of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation
10. objective evidence indicating previous or concurrent pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, radiation-induced pneumonia, drug-related pneumonia, severe impairment of lung function, etc
11. patients with hypertension that cannot be restored to the normal range (systolic blood pressure ≤ 140 mmHg / diastolic blood pressure ≤ 90 mmHg) after treatment with antihypertensive drugs for 3 months
12. patients with uncontrolled clinical symptoms or diseases of the heart, including but not limited to congestive heart failure (NYHA grade > II); unstable or severe angina; acute myocardial infarction within 6 months; patients with clinically significant supraventricular or ventricular arrhythmia requiring clinical intervention; left ventricular ejection fraction (LVEF) < 50%
13. patients at risk of serious bleeding, including but not limited to severe bleeding (bleeding > 30 ml within 3 months), hemoptysis (bleeding > 5 ml within 4 weeks), and thromboembolism events (within the past 12 months)
14. with symptoms indicating Grade 2+ peripheral neuropathy
15. participating in other clinical trials, or participating in any clinical study for drugs within previous 4 weeks
16. other situations that the researchers regard as not suitable for inclusion.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-03-01 (Estimated); Primary Completion 2023-02-28 (Estimated); Study Completion 2023-02-28 (Estimated)

PRIMARY OUTCOMES:
R0 resection rate | 3 years
  proportion of patients for whom radical resection can be achieved

SECONDARY OUTCOMES:
ORR | 3 years
  objective response rate
DFS | 3 years
  disease free survival (period)
3-year DFS | 3 years
  3-year disease free survival (rate)
PFS | 3 years
  progression free survival (period)
OS | 3 years
  overall survival (period)
1-year OS | 1 year
  1-year overall survival (rate)
3-year OS | 3 years
  3-year overall survival (rate)

CONTACTS AND LOCATIONS:
Overall Officials: Wei Deng, Study Director — Beijing Friendship Hospital
Locations (1):
- Beijing Friendship Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided